CLINICAL TRIAL: NCT02319265
Title: Dose Assessment of Melatonin in Sepsis Trial
Acronym: DAMSEL2
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study registered elsewhere and is not covered by FDA
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3/035/14
Record Dates: First submitted 2014-12-03; First posted 2014-12-18 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Sepsis
Keywords: sepsis; antioxidant; melatonin; inflammation
MeSH Terms: conditions — Sepsis; Inflammation | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Melatonin at a dose of either 50mg (50ml) or 100mg (100ml) to be decided after an initial PK study to be given at intervals to be decided after PK data is available, for 72h. Oral liquid via nasogastric tube.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo at a dose of either 50ml or 100ml (to be decided after an initial PK study) to be given at intervals to be decided after PK data, is available for 72h. Oral liquid via nasogastric tube.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Oral liquid
  Other Names: N-acetyl-5-methoxytryptamine

SUMMARY:
DAMSEL 2 is a pilot Phase II study in patients with sepsis. Stage 1 will assess the pharmacokinetics of melatonin and its major metabolite after a single dose of 50 or 100mg exogenous melatonin in two small groups of patients with sepsis in order to make dosing and dosing interval decisions for Stage 2.

Stage 2 is a double blind randomised controlled trial of melatonin in patients with sepsis at the dose and dosing interval decided after Stage 1. Measurements of melatonin and its major metabolite, and an array of biomarkers of inflammation and oxidative stress will be made, plus transcriptome (mRNA) analysis. This study will inform a planned larger phase II trial.

DETAILED DESCRIPTION:
Antioxidant therapy targeted at mitochondria has the potential to reduce inflammation, mitochondrial damage and organ dysfunction in sepsis. Melatonin accumulates in mitochondria and both it and its metabolites have potent antioxidant and anti-inflammatory activity, preventing organ dysfunction in a rat model of sepsis. In a recent Phase I dose escalation study (DAMSEL 1) the investigators showed that oral doses of melatonin in healthy subjects were well tolerated with no adverse events and resulted in levels of circulating melatonin and its major metabolite which had beneficial anti-inflammatory and antioxidant actions in ex vivo studiesStage 1 will assess the pharmacokinetics of melatonin and its major metabolite after a single dose of 50 or 100mg exogenous melatonin in two small groups of patients with sepsis in order to make dosing and dosing interval decisions for Stage 2.

Stage 2 is a double blind randomised controlled trial of melatonin in patients with sepsis at the dose and dosing interval decided after Stage 1. Measurements of melatonin and its major metabolite, and an array of biomarkers of inflammation and oxidative stress will be made, plus transcriptome (mRNA) analysis. This study will inform a planned larger phase II trial.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (16 years or over) on the ICU at Aberdeen Royal Infirmary with sepsis due to community acquired pneumonia who are within 24h of fulfilling the criteria for sepsis with clinical suspicion of pneumonia and the presence of chest X-ray changes consistent with pneumonia will be recruited. The criteria for sepsis are:

* clinical suspicion or evidence of acute infection
* systemic inflammatory response syndrome, defined by two or more of the following:

  1. Core temperature <36 or >38°C;
  2. tachycardia: heart rate > 90 beats/min;
  3. tachypnoea: respiratory rate > 20 breaths/min or ventilated;
  4. leucocyte count >12 x 109/L or <4 x 109/L.

Exclusion Criteria:

* <16 years old,
* have a life expectancy <24h,
* have metastatic cancer or immunosuppression,
* are receiving steroids (>20mg/d prednisolone or equivalent, used regularly for >2 weeks prior to ICU admission)
* women of child bearing potential without a negative pregnancy test or a history of surgical sterilization.
* patients receiving fluvoxamine or nifedipine,
* have overt hepatic failure
* unable to tolerate oral medication
* known to be hypersensitive to trial medication and/or excipients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Completion of enrollment of 10 patients to Stage 1 | 6 months
  Stage 1= first 5 patients 50mg, second 5 patients 100mg oral melatonin liquid, open label

SECONDARY OUTCOMES:
Composite pharmacokinetic measures for each dose in Stage 1 (T max, CMax and AUC) | 6 months
  T max, CMax and AUC of melatonin and 6-hydroxymelatonin sulphate levels at two doses of melatonin.
Composite biomarker measures in Stage 2 ( linear discriminant analysis, hierarchical regression and hierarchical cluster analysis) | 2 years
  Multiplex biomarker analysis will be used; linear discriminant analysis, hierarchical regression and hierarchical cluster analysis will be used to explore relationships between biomarkers
28d all cause mortality in Stage 2 | 2 years
  Survival status at 28d
Arterial blood lactate (stage 1 and stage 2) | 2 years
  Absolute arterial lactate measures at various time points; change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Galley, Study Director — Univetsity of Aberdeen
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No